CLINICAL TRIAL: NCT04016792
Title: An Analog Classroom Study: Efficacy and Safety of SPN-812 in Children With Attention-Deficit/Hyperactivity Disorder
Brief Title: Classroom Study of SPN-812 in Children With ADHD
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped before enrollment due to non-safety related corporate decision.
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 812P308
Record Dates: First submitted 2019-07-10; First posted 2019-07-11 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo qd
  Interventions: Drug: Placebo
- SPN-812 (Experimental): 200 mg SPN-812
  Interventions: Drug: 200 mg SPN-812

INTERVENTIONS:
Drug: Placebo — Placebo will be administered once daily
  Other Names: PBO
  Arms: Placebo
Drug: 200 mg SPN-812 — 200 mg SPN-812 will be administered once daily and compared to Placebo
  Other Names: SPN-812 Fixed Dose
  Arms: SPN-812

SUMMARY:
This study will evaluate the efficacy and safety of SPN-812, an extended-release formulation of viloxazine, compared to placebo in children in an analog classroom setting.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled, parallel-group, 2-arm, analog classroom study to evaluate the efficacy and safety of 200 mg/day SPN-812 compared to placebo in the treatment of children aged 6 through 11 years with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, 6 to <12 years of age at screening.
2. Primary diagnosis of ADHD (inattentive, hyperactive, or combined presentation) or ADHD with comorbidity of mild to moderate oppositional defiant disorder (ODD) according to the DSM-5, confirmed with the MINI-KID at screening.
3. ADHD-RS-5 (Home Version: Child, Investigator Administered and Scored) score ≥28 at screening and at baseline (can be assessed 1 to 2 days before Visit 3).
4. CGI-S score ≥ 4 at baseline (can be assessed 1 to 2 days before Visit 3).
5. Body weight ≥ 20 kg.
6. Free of medication for the treatment of ADHD for at least 1 week prior to randomization and agreement to remain so throughout participation in the study.
7. Have the ability to complete PERMP assessments by qualifying for at least the Basic level at screening (see Section 6.1.2).
8. Considered medically healthy by the Investigator via assessment of physical examination, medical and psychiatric histories, clinical laboratory tests, vital signs, and ECG.
9. Written informed consent obtained from the subject's parent or legal representative, and written informed assent (if applicable) obtained from the subject.
10. Subject and parent(s)/legal guardian(s) are willing and able to comply with all of the procedures and requirements defined in the protocol, including parents(s)/legal guardian(s) oversight of the morning dosing of SM.
11. Subject has lived with the same parent(s)/legal guardian(s) for > 6 months.
12. FOCP must be either sexually inactive (abstinent) or, if sexually active, must agree to use one of the following highly effective contraceptive methods beginning 30 days prior to the first dose, throughout their participation in the study:

    1. Simultaneous use of male condom and intra-uterine contraceptive device placed at least 4 weeks prior to the first SM administration;
    2. Surgically sterile male partner;
    3. Simultaneous use of male condom and diaphragm with spermicide;
    4. Established hormonal contraceptive.

Exclusion Criteria:

1. Current diagnosis of major psychiatric disorders or intellectual disabilities are excluded, including severe ODD, conduct disorder, autism spectrum disorders, simple phobias, or learning disorders. Subjects with a history of Major Depressive Disorder are eligible if the subject has not experienced an episode or required pharmacotherapy within the 6 months prior to the screening visit.
2. Current diagnosis of major neurological disorders. Subjects with seizures or a history of seizure disorder within the immediate family (siblings, parents). Febrile seizures are not exclusionary and will be assessed on a case-by-case basis. If for any reason the subject received medication for a febrile seizure, this it will be exclusionary.
3. Subject has failed two treatment courses (dose and duration) of stimulant or nonstimulant for ADHD; subjects who are treatment naïve are not excluded from participating.
4. In the opinion of the investigator, current diagnosis of significant systemic disease.
5. Body mass index greater than 95th percentile for the appropriate age and gender.
6. At screening, uncontrolled thyroid disorder defined as thyroid stimulating hormone ≤ 0.8 x the lower limit of normal or ≥ 1.25 x the upper limit of normal for the reference laboratory.
7. Any clinically significant abnormal laboratory test, urine test, ECG result, or physical exam finding that, in the opinion of the Investigator, would interfere with the safety of the subject.
8. Evidence of suicidality (defined as either active suicidal plan/intent or active suicidal thoughts within the year prior to screening visit, or a lifetime suicide attempt).
9. History of an allergic reaction to viloxazine or its excipients.
10. Any food allergy, intolerance, restriction or special diet that, in the opinion of the Investigator, could contraindicate the subject's participation in this study.
11. Subjects who received any investigational drug within the longer of 30 days or 5 half-lives prior to Day 2 dosing of SM.
12. Subjects who participated in previous SPN-812 clinical trials.
13. Subjects who have participated in another analog classroom study within 6 months prior to screening visit and subjects who have participated in more than one classroom study.
14. Positive urine drug screen at screening visit. A positive test for amphetamines is not exclusionary for subjects receiving a stimulant ADHD medication at the time of the screening visit, however, an additional urine drug screen should be performed at Visit 3. Subjects must discontinue all prohibited/ADHD medication (including stimulant, clonidine and guanfacine) at least 7 days prior to Visit 3.
15. Pregnancy, breastfeeding, or refusal to practice abstinence or acceptable birth control during the study (for FOCP).
16. Any reason that, in the opinion of the Investigator, would prevent the subject from participating in the study.
17. Subjects currently taking specific concomitant medications known to be CYP1A2 substrates (e.g., theophylline, melatonin, olanzapine, duloxetine).

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy of SPN-812 assessed by Swanson, Kotkin, Agler, M-Flynn, and Pelham Scale- Combined Score (SKAMP-CS) | 29 days
  Change from baseline in mean SKAMP-CS, averaged from 8 post-dose assessments collected across the 12-h analog classroom day

SECONDARY OUTCOMES:
Effect of SPN-812 assessed longitudinally by SKAMP-CS | 29 days
  Change from baseline in SKAMP-CS at individual time points across the classroom day
Effect of SPN-812 assessed longitudinally by Permanent Product (PERMP) math test | 29 days
  Change from baseline in PERMP math test number attempted and number correct at individual time points across the classroom day
Effect of SPN-812 on Clinical Global Impression-Severity (CGI-S) scale | 29 days
  Change from baseline in CGI-S score
Effect of SPN-812 on SKAMP Attention and SKAMP Deportment subscales | 29 days
  Change from baseline in mean SKAMP Attention and SKAMP Deportment scores, averaged from 8 post-dose assessments
Effect of SPN-812 assessed longitudinally on SKAMP Attention and SKAMP Deportment subscales | 29 days
  Change from baseline in SKAMP Attention and SKAMP Deportment scores at individual time points across the classroom day
Effect of SPN-812 assessed by ADHD Rating Scale-5 (ADHD-RS-5) Total Score and subscales | 29 days
  Change from baseline in ADHD-RS-5 Total Score, Hyperactivity/Impulsivity score and Inattention score
Effect of SPN-812 assessed by Clinical Global Impression-Improvement (CGI-I) scale | 29 days
  Change from baseline in CGI-I score
Effect of SPN-812 assessed by categorical CGI-I Responder Rate | 29 days
  Change from baseline in categorical CGI-I score
Effect of SPN-812 assessed by 50% Responder Rate to ADHD Rating Scale-5 baseline | 29 days
  Percentage of subjects with at least 50% reduction in ADHD-RS-5 total score
Effect of SPN-812 assessed by Conners 3rd Edition-Parent Report Short Form (Conners 3-PS) Composite T score | 29 days
  Change from baseline in Conners 3-PS Composite T score

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schwabe, MD, Study Director — Chief Medical Officer

IPD SHARING:
Plan to Share IPD: No